CLINICAL TRIAL: NCT06926322
Title: Nano-based Medicaments Versus Double Antibiotic Paste in Managing Non-vital Primary Molars: A Randomized Clinical Trial and In-Vitro Study
Brief Title: Evaluation of Different Medicaments in the Management of Necrotic Primary Molars by Lesion Sterilization and Tissue Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Ehab Abdel Razik Kamel, Assistant Lecturer of Pediatric Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED-25-D1
Record Dates: First submitted 2025-04-05; First posted 2025-04-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pain, Postoperative; Root Resorption; Persistent Infection; Necrotic Pulp
MeSH Terms: conditions — Pain, Postoperative; Root Resorption; Persistent Infection; Dental Pulp Necrosis | interventions — Ciprofloxacin; Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The current study will be a triple-blind study. The participants will be blind to the study groups they will be assigned to. The evaluators will also be blind to the study groups during clinical and radiographic examination. The operator will not be blind to the study groups because of the difference between the used medicaments. The statistician will be unaware of the study group's allocation during statistical analysis of the data collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional double antibiotic paste (Active Comparator): After local anesthesia administration and rubber dam isolation, access cavity will be performed and the studied medicament will be placed onto the floor of the pulp chamber. Teeth will be finally restored with stainless steel crowns in the same visit.
  Interventions: Drug: Conventional double antibiotic paste of Metronidazole 500 mg plus Ciprofloxacin 500 mg mixed with propylene glycol
- double antibiotic paste-loaded chitosan-coated silver nanoparticles (Experimental): After local anesthesia administration and rubber dam isolation, access cavity will be performed and the studied medicament will be placed onto the floor of the pulp chamber. Teeth will be finally restored with stainless steel crowns in the same visit.
  Interventions: Drug: Double antibiotic paste of Metronidazole and Ciprofloxacin loaded chitosan-coated silver nanoparticles
- chitosan-coated silver nanoparticles (Experimental): After local anesthesia administration and rubber dam isolation, access cavity will be performed and the studied medicament will be placed onto the floor of the pulp chamber. Teeth will be finally restored with stainless steel crowns in the same visit.
  Interventions: Drug: chitosan-coated silver nanoparticles

INTERVENTIONS:
Drug: Conventional double antibiotic paste of Metronidazole 500 mg plus Ciprofloxacin 500 mg mixed with propylene glycol — The studied medicament will be placed onto the floor of the pulp chamber.
  Arms: Conventional double antibiotic paste
Drug: Double antibiotic paste of Metronidazole and Ciprofloxacin loaded chitosan-coated silver nanoparticles — The studied medicament will be placed onto the floor of the pulp chamber.
  Arms: double antibiotic paste-loaded chitosan-coated silver nanoparticles
Drug: chitosan-coated silver nanoparticles — The studied medicament will be placed onto the floor of the pulp chamber.
  Arms: chitosan-coated silver nanoparticles

SUMMARY:
Management of non-vital primary molars is challenging due to the natural anatomy of primary teeth, patients' young age, and their behavior toward dental treatment. A simple and effective technique such as Lesion Sterilization and Tissue Repair offers a solution to cases with poor prognosis; however, the medicaments used in this technique have some limitations. This study will evaluate three different medicaments regarding the clinical success, radiographic success, and antibacterial activity.

DETAILED DESCRIPTION:
This randomized controlled trial will include 108 non-vital mandibular primary molars in children aged 4-8. Patients will be randomly allocated into three groups according to the studied medicaments as one positive control group and two experimental groups. The groups are as follows:

Group I (conventional double antibiotic paste) positive control group Group II (double antibiotic paste-loaded chitosan-coated silver nanoparticles) experimental group Group III (chitosan-coated silver nanoparticles) experimental group

The antibacterial activity of studied medicaments will be tested against Enterococcus Faecalis bacteria in planktonic and biofilm forms. Teeth will be evaluated clinically and radiographically to obtain baseline data. After local anesthesia administration and isolation of teeth, an access cavity will be performed, then the medicament will be placed over the floor of the pulp chamber according to the corresponding group. Afterwards, teeth will be filled with resin-modified zinc oxide and eugenol followed by stainless steel crowns. Blinded clinical evaluation will be done at baseline, 1, 6, and 12 months and blinded radiographic evaluation will be done at baseline, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cooperative children of both sexes in the age range of 4-8 years old.
* Children with consenting parents who accept to participate in the study and sign the consent forms.
* Children with mandibular primary molars with clinical and radiographic signs of pulpal necrosis.

Exclusion Criteria:

* Children with hypersensitivity to any of the used medicaments.
* Non-restorable teeth without sufficient coronal structure for placement of rubber dam isolation and restoration with stainless steel crowns
* Non-restorable teeth with perforated pulpal floor

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1,6, and 12 months follow up
  1. Absence/decrease of pain related to the treated teeth including patient reported pain or sensitivity to palpation/percussion
  2. Absence/decrease of gingival swelling related to the treated teeth
  3. Absence/decrease of pathological mobility related to the treated teeth
Radiographic success | 6 and 12 months follow up
  1. Absence/decrease/stasis of furcation radiolucency related to the treated teeth
  2. Absence/stasis of pathological root resorption of the treated teeth

SECONDARY OUTCOMES:
Antibacterial activity of studied medicaments against Enterococcus Faecalis bacteria | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Khattab, Study Director — Ain Shams University
Locations (1):
- Faculty of dentistry Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided